CLINICAL TRIAL: NCT05202210
Title: Constitution of a Biological Collection to Study the Pathophysiology in Noonan Syndrome and to Identify Predictive Factors of Disease Progression
Brief Title: Constitution of a Biological Collection to Study the Pathophysiology in Noonan Syndrome
Acronym: Noonan
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/21/0361
Record Dates: First submitted 2022-01-07; First posted 2022-01-21 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Noonan Syndrome
Keywords: Biological collection; Noonan Syndrome
MeSH Terms: conditions — Noonan Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with Noonan syndrome: extra sample of blood and urine will be collected and stored for research utilisation
  Interventions: Biological: blood and urine sampling

INTERVENTIONS:
Biological: blood and urine sampling — extra sample of blood and urine will be collected

SUMMARY:
The present study will establish a collection of biological samples from Noonan patients to be used for research purposes only, with due respect for confidentiality.

DETAILED DESCRIPTION:
Noonan syndrome is a rare autosomal dominant genetic disorder characterized by a combination of typical facial features, heart defects, short stature, skeletal abnormalities, mild developmental delay and a predisposition to myeloproliferative disorders. This syndrome is caused by germline mutations in genes encoding components or regulators of the Rat Sarcoma (RAS) / extracellular signal-regulated kinase (ERK) signaling pathway, which is essential for cell cycle differentiation, growth, and senescence.

Patients with Noonan syndrome or related diseases are followed at the children's hospital, Toulouse University Hospital. During regular check-up visits, an extra sample of blood and urine will be collected and stored for research utilisation with the patient's consent. The ultimate objective of this collection is to provide available biological resources to facilitate the development of subsequent studies aimed at better characterizing the multisystemic disorders in Noonan syndrome, to understand the pathophysiology of the disease, and to identify biological factors that predict the severity and progression of the disease. The possibility of having systematically collected biological resources will make it possible to answer certain questions more quickly depending on the progress of research.

ELIGIBILITY:
Inclusion Criteria:

* Children aged at least 3 years old or adult with Noonan syndrome
* Patients affiliated to or beneficiaries of a social security scheme
* Patients able to receive information on the progress of the study and understand the information form to participate in the study. That implies to master the French language and not to be subject to a restriction of rights by the judicial authorities
* Patients or legal representative who have given their consent to participate in the study (expression of no objection)

Exclusion Criteria:

* Patients subject to a legal protection measure (guardianship, curators, or safeguard of justice)
* Pregnant or breastfeeding women

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Noonan syndrome
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-26 (Actual); Primary Completion 2027-01-26 (Estimated); Study Completion 2032-01-26 (Estimated)

PRIMARY OUTCOMES:
Constitution of a biological collection from patients with Noonan or related syndromes. | inclusion
  extra sample of blood and urine will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Thomas EDOUARD, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Purpan University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No